CLINICAL TRIAL: NCT04448756
Title: A Phase II, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of M5049 in Hospitalized Participants With COVID-19 Pneumonia (ANEMONE)
Brief Title: Study of M5049 in Participants With COVID-19 Pneumonia (ANEMONE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS200569_0026; 2020-002248-22 (EudraCT Number)
Record Dates: First submitted 2020-06-25; First posted 2020-06-26 (Actual); Results first posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-05

CONDITIONS: Coronavirus Disease 2019
Keywords: COVID-19; Severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- M5049 50 mg (Experimental)
  Interventions: Drug: M5049
- M5049 100 mg (Experimental)
  Interventions: Drug: M5049
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: M5049 — Participants received M5049 50 milligram (mg) orally twice daily for 14 days.
  Arms: M5049 50 mg
Drug: M5049 — Participants received M5049 100 mg orally twice daily for 14 days.
  Arms: M5049 100 mg
Drug: Placebo — Participants received placebo tablets matched to M5049 daily for 14 days.
  Arms: Placebo

SUMMARY:
The study will evaluate the safety and efficacy of orally-administered M5049 in Coronavirus disease 2019 (COVID-19) pneumonia participants who are hospitalized but not on mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Participant provides signed informed consent prior to the initiation of any study assessments
* Has laboratory-confirmed SARS-CoV-2 Infection as determined by nucleic acid amplification test, polymerase chain reaction, antigen test or other commercial or public health assay (based on locally acceptable accepted guidelines) in a sample collected less than (<)10 days prior to randomization
* Has chest imaging consistent with COVID-19 pneumonia (as per locally accepted guidelines) If chest imaging is not available during Screening, please discuss with Medical Monitor or designee regarding evidence of probable COVID-19 pneumonia for study participant eligibility
* Not on mechanical ventilation or ECMO
* Has an SpO2 less than (<) 94 percent in room air And able to maintain a partial pressure of oxygen (PaO2)/fraction of inspired oxygen (FiO2) greater than or equal to (>=) 150 (Or equivalent SpO2/FiO2 >=190) with a maximum FiO2 0.4 if participant is on chronic low oxygen therapy (less than or equal to 2 Liter), assess their current baseline oxygen requirements for eligibility
* Requires hospitalization
* Other protocol defined inclusion criteria may apply

Exclusion Criteria:

* Any condition that could interfere with the study objectives, conduct or evaluation in the opinion of the Investigator or Sponsor or designee
* Significantly uncontrolled medical illness (eg, cardiovascular disease, hypertension, diabetes mellitus, obstructive lung disease, neurological associated with seizures (example: cerebrovascular accident/stroke, acute brain infection, traumatic brain injury, progressive brain disease, congenital brain disease or neuropsychiatric disorder)
* Known active infection other than COVID-19
* Pregnancy or Breastfeeding
* Other protocol defined exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (21):
- United States (5):
  - LAC-USC Medical Center, Los Angeles, California
  - Sharp Chula Vista Medical Center, San Diego, California
  - Henry Ford Medical Center, Detroit, Michigan
  - Holy Name Hospital - Dept of Multiple Sclerosis Comp Care Center, Teaneck, New Jersey
  - Christus Spohn Hospital Corpus Christi-Memorial, Corpus Christi, Texas
- Brazil (10):
  - Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte
  - Hospital Dia do Pulmão, Blumenau
  - Hospital São José - Sociedade Literária e Caritativa Santo Agostinho, Criciúma
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - HMCG - Hospital e Maternidade Dr. Christovão da Gama, Santo André
  - Pesquisare, Santo André
  - Hospital Alemão Oswaldo Cruz, São Paulo
  - Hospital Bandeirantes / Hospital Leforte Liberdade, São Paulo
  - Hospital Leforte Morumbi, São Paulo
  - Instituto de Infectologia Emílio Ribas, São Paulo
- Philippines (6):
  - Manila Doctors Hospital, Manila
  - Medical Center Manila - Medicine, Manila
  - Lung Center of the Philippines - Medicine, Quezon
  - Quirino Memorial Medical Center, Quezon
  - Veterans Memorial Medical Center, Quezon
  - East Avenue Medical Center, Quezon City

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- [Derived] McKinnon JE, Santiaguel J, Murta de Oliveira C, Yu D, Khursheed M, Moreau F, Klopp-Schulze L, Shaw J, Roy S, Kao AH; ANEMONE Study Team. Enpatoran in COVID-19 pneumonia: Safety and efficacy results from a phase II randomized trial. Clin Transl Sci. 2023 Dec;16(12):2640-2653. doi: 10.1111/cts.13658. Epub 2023 Oct 23. PMID 37873555
- [Derived] Klopp-Schulze L, Shaw JV, Dong JQ, Khandelwal A, Vazquez-Mateo C, Goteti K. Applying Modeling and Simulations for Rational Dose Selection of Novel Toll-Like Receptor 7/8 Inhibitor Enpatoran for Indications of High Medical Need. Clin Pharmacol Ther. 2022 Aug;112(2):297-306. doi: 10.1002/cpt.2606. Epub 2022 May 21. PMID 35390178
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200569_0026
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 200 participants were screened for this study. Of which, 149 participants were randomized into the study.
Groups:
- Placebo: Participants received matched placebo tablets to M5049 daily for 14 days.
- M5049 50 Milligram (mg): Participants received M5049 50 milligram (mg) orally twice daily for 14 days.
- M5049 100 mg: Participants received M5049 100 mg orally twice daily for 14 days.
Period: Overall Study
Arm/Group | Placebo | M5049 50 Milligram (mg) | M5049 100 mg
Started | 49 | 54 | 46
Completed | 46 | 49 | 45
Not Completed | 3 | 5 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Participant unable to attend Day 60 visit | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 1
Not completed — Death | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who had received at least one dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | M5049 50 Milligram (mg) | M5049 100 mg | Total
Number analyzed (Participants) | 49 | 54 | 46 | 149
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.4 (14.09) | 51.0 (12.25) | 49.2 (12.35) | 49.6 (12.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 14 | 51
  Male | 31 | 35 | 32 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 38 | 29 | 96
  Not Hispanic or Latino | 20 | 15 | 15 | 50
  Unknown or Not Reported | 0 | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 13 | 16 | 12 | 41
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 3 | 7 | 4 | 14
  White | 22 | 20 | 25 | 67
  More than one race | 6 | 7 | 0 | 13
  Unknown or Not Reported | 4 | 4 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Time to Recovery
Description: Time to recovery was defined as the time from first dose (Day 1) to first occurrence of World Health Organization (WHO) 9-point ordinal scale 3 or less. The scoring is assessed with the following ordinal scale: 0. Uninfected: no clinical or virological evidence of infection; 1. Ambulatory: no limitation of activities; 2. Ambulatory: limitation of activities; 3. Hospitalized, mild disease: hospitalized, no oxygen therapy; 4. Hospitalized, mild disease: oxygen by mask or nasal prongs; 5. Hospitalized, severe disease: noninvasive ventilation or high-flow oxygen; 6. Hospitalized, severe disease: intubation and mechanical ventilation; 7. Hospitalized, severe disease: ventilation plus additional organ support for example: vasopressors or Extracorporeal membrane oxygenation (ECMO); 8. Death.
Time Frame: Day 1 through Day 28
Population: Intent-to-Treat analysis set included all participants who had received at least one dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | M5049 50 Milligram (mg) | M5049 100 mg
Number analyzed (Participants) | 49 | 54 | 46
Days | 3.4 [2.7 to 4.9] | 3.7 [2.6 to 4.0] | 3.9 [2.0 to 4.8]

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Adverse Events of Special Interests (AESIs), TEAEs Leading to Treatment Discontinuation and Serious TEAEs (SAEs) According to NCI-CTCAE Version 5.0
Description: Adverse Event (AE) was defined any untoward medical occurrence in a participant administered with a study drug, which does not necessarily had a causal relationship with this treatment. Serious AE was defined AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs: TEAEs was defined as events with onset date or worsening during the on treatment period. TEAEs included serious TEAEs and non-serious TEAEs.
Time Frame: Day 1 through Day 60
Population: Safety analysis set included all participants who had received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | M5049 50 Milligram (mg) | M5049 100 mg
Number analyzed (Participants) | 49 | 54 | 46
Participants
  Participants with any TEAE | 28 | 34 | 26
  Participants with any AESIs | 2 | 2 | 0
  Participants with TEAEs leading to discontinuation | 4 | 4 | 1
  Participants with Serious TEAEs | 9 | 5 | 1

3. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Parameters
Description: Laboratory investigation included hematology and biochemistry. The number of participants with clinically significant changes from baseline in laboratory parameters were reported. Clinical significance was determined by the investigator.
Time Frame: Day 1 through Day 28
Population: Safety analysis set included all participants who had received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | M5049 50 Milligram (mg) | M5049 100 mg
Number analyzed (Participants) | 49 | 54 | 46
Participants | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in 12-Lead Electrocardiogram (ECG) Measurements
Description: 12-lead ECG recordings included rhythm, heart rate (as measured by RR interval), PR interval, QRS duration, and QT interval. 12-lead ECG recordings were obtained after the participants have rested for at least 10 minutes in semisupine position. Clinical significance was determined by the investigator. The number of participants with clinically significant changes from baseline in 12-lead ECG findings were reported.
Time Frame: Day 1 through Day 28
Population: Safety analysis set included all participants who had received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | M5049 50 Milligram (mg) | M5049 100 mg
Number analyzed (Participants) | 49 | 54 | 46
Participants | 1 | 0 | 0

5. Secondary Outcome: Percentage of Participants Alive and Not Requiring Supplemental Oxygenation
Description: The percentage of participants who were alive and did not require supplemental oxygenation or ventilatory support (including noninvasive or mechanical ventilation and Extra Corporeal Membrane Oxygenation [ECMO]) reported.
Time Frame: Day 3, Day 7, Day 14, Day 21 and Day 28
Population: Intent-to-Treat analysis set included all participants who had received at least one dose of study intervention. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signified those participants who were evaluable for the specified category at given time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | M5049 50 Milligram (mg) | M5049 100 mg
Number analyzed (Participants) | 49 | 51 | 44
Percentage of participants
  At Day 3 | 30.6 [19.5 to 44.5] | 27.5 [17.1 to 40.9] | 38.6 [25.7 to 53.4]
  At Day 7: number analyzed (Participants) | 47 | 48 | 42
  At Day 7 | 76.6 [62.8 to 86.4] | 83.3 [70.4 to 91.3] | 83.3 [69.4 to 91.7]
  At Day 14: number analyzed (Participants) | 48 | 49 | 44
  At Day 14 | 89.6 [77.8 to 95.5] | 89.8 [78.2 to 95.6] | 100.0 [92.0 to 100.0]
  At Day 21: number analyzed (Participants) | 43 | 48 | 43
  At Day 21 | 93.0 [81.4 to 97.6] | 93.8 [83.2 to 97.9] | 100.0 [91.8 to 100.0]
  At Day 28: number analyzed (Participants) | 48 | 51 | 44
  At Day 28 | 93.8 [83.2 to 97.9] | 98.0 [89.7 to 99.7] | 97.7 [88.2 to 99.6]

6. Secondary Outcome: Number of Participants in Each Clinical Status Category Based on 9-Point Ordinal Scale
Description: Clinical status was based on data collected on the 'Ordinal Scale for Clinical Status and is assessed with the following ordinal scale: 0. Uninfected: no clinical or virological evidence of infection; 1. Ambulatory: no limitation of activities; 2. Ambulatory: limitation of activities; 3. Hospitalized, mild disease: hospitalized, no oxygen therapy; 4. Hospitalized, mild disease: oxygen by mask or nasal prongs; 5. Hospitalized, severe disease: noninvasive ventilation or high-flow oxygen; 6. Hospitalized, severe disease: intubation and mechanical ventilation; 7. Hospitalized, severe disease: ventilation plus additional organ support for example: vasopressors or ECMO; 8. Death.
Time Frame: Baseline, Day 2, Day 3, Day 4, Day 5, Day 7, Day 10, Day 14, Day 21, Day 28, Day 44, Day 60
Population: Intent-to-Treat analysis set included all participants who had received at least one dose of study intervention. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and Number Analyzed" signified those participants who were evaluable for the specified category at given time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | M5049 50 Milligram (mg) | M5049 100 mg
Number analyzed (Participants) | 49 | 53 | 46
Participants
  Participants with Scale 0 at Baseline: number analyzed (Participants) | 49 | 52 | 44
  Participants with Scale 0 at Baseline | 0 | 0 | 0
  Participants with Scale 1 at Baseline: number analyzed (Participants) | 49 | 52 | 44
  Participants with Scale 1 at Baseline | 0 | 0 | 0
  Participants with Scale 2 at Baseline: number analyzed (Participants) | 49 | 52 | 44
  Participants with Scale 2 at Baseline | 0 | 0 | 0
  Participants with Scale 3 at Baseline: number analyzed (Participants) | 49 | 52 | 44
  Participants with Scale 3 at Baseline | 1 | 0 | 0
  Participants with Scale 4 at Baseline: number analyzed (Participants) | 49 | 52 | 44
  Participants with Scale 4 at Baseline | 48 | 52 | 44
  Participants with Scale 5 at Baseline: number analyzed (Participants) | 49 | 52 | 44
  Participants with Scale 5 at Baseline | 0 | 0 | 0
  Participants with Scale 6 at Baseline: number analyzed (Participants) | 49 | 52 | 44
  Participants with Scale 6 at Baseline | 0 | 0 | 0
  Participants with Scale 7 at Baseline: number analyzed (Participants) | 49 | 52 | 44
  Participants with Scale 7 at Baseline | 0 | 0 | 0
  Participants with Scale 8 at Baseline: number analyzed (Participants) | 49 | 52 | 44
  Participants with Scale 8 at Baseline | 0 | 0 | 0
  Participants with Scale 0 at Day 2: number analyzed (Participants) | 48 | 53 | 46
  Participants with Scale 0 at Day 2 | 0 | 0 | 0
  Participants with Scale 1 at Day 2: number analyzed (Participants) | 48 | 53 | 46
  Participants with Scale 1 at Day 2 | 1 | 0 | 0
  Participants with Scale 2 at Day 2: number analyzed (Participants) | 48 | 53 | 46
  Participants with Scale 2 at Day 2 | 0 | 1 | 2
  Participants with Scale 3 at Day 2: number analyzed (Participants) | 48 | 53 | 46
  Participants with Scale 3 at Day 2 | 9 | 12 | 13
  Participants with Scale 4 at Day 2: number analyzed (Participants) | 48 | 53 | 46
  Participants with Scale 4 at Day 2 | 35 | 39 | 30
  Participants with Scale 5 at Day 2: number analyzed (Participants) | 48 | 53 | 46
  Participants with Scale 5 at Day 2 | 3 | 0 | 1
  Participants with Scale 6 at Day 2: number analyzed (Participants) | 48 | 53 | 46
  Participants with Scale 6 at Day 2 | 0 | 1 | 0
  Participants with Scale 7 at Day 2: number analyzed (Participants) | 48 | 53 | 46
  Participants with Scale 7 at Day 2 | 0 | 0 | 0
  Participants with Scale 8 at Day 2: number analyzed (Participants) | 48 | 53 | 46
  Participants with Scale 8 at Day 2 | 0 | 0 | 0
  Participants with Scale 0 at Day 3: number analyzed (Participants) | 49 | 51 | 44
  Participants with Scale 0 at Day 3 | 0 | 0 | 0
  Participants with Scale 1 at Day 3: number analyzed (Participants) | 49 | 51 | 44
  Participants with Scale 1 at Day 3 | 2 | 2 | 1
  Participants with Scale 2 at Day 3: number analyzed (Participants) | 49 | 51 | 44
  Participants with Scale 2 at Day 3 | 1 | 3 | 2
  Participants with Scale 3 at Day 3: number analyzed (Participants) | 49 | 51 | 44
  Participants with Scale 3 at Day 3 | 12 | 9 | 14
  Participants with Scale 4 at Day 3: number analyzed (Participants) | 49 | 51 | 44
  Participants with Scale 4 at Day 3 | 29 | 36 | 26
  Participants with Scale 5 at Day 3: number analyzed (Participants) | 49 | 51 | 44
  Participants with Scale 5 at Day 3 | 4 | 0 | 1
  Participants with Scale 6 at Day 3: number analyzed (Participants) | 49 | 51 | 44
  Participants with Scale 6 at Day 3 | 1 | 1 | 0
  Participants with Scale 7 at Day 3: number analyzed (Participants) | 49 | 51 | 44
  Participants with Scale 7 at Day 3 | 0 | 0 | 0
  Participants with Scale 8 at Day 3: number analyzed (Participants) | 49 | 51 | 44
  Participants with Scale 8 at Day 3 | 0 | 0 | 0
  Participants with Scale 0 at Day 4: number analyzed (Participants) | 37 | 42 | 32
  Participants with Scale 0 at Day 4 | 0 | 0 | 0
  Participants with Scale 1 at Day 4: number analyzed (Participants) | 37 | 42 | 32
  Participants with Scale 1 at Day 4 | 0 | 1 | 0
  Participants with Scale 2 at Day 4: number analyzed (Participants) | 37 | 42 | 32
  Participants with Scale 2 at Day 4 | 0 | 1 | 0
  Participants with Scale 3 at Day 4: number analyzed (Participants) | 37 | 42 | 32
  Participants with Scale 3 at Day 4 | 14 | 16 | 11
  Participants with Scale 4 at Day 4: number analyzed (Participants) | 37 | 42 | 32
  Participants with Scale 4 at Day 4 | 17 | 22 | 21
  Participants with Scale 5 at Day 4: number analyzed (Participants) | 37 | 42 | 32
  Participants with Scale 5 at Day 4 | 5 | 1 | 0
  Participants with Scale 6 at Day 4: number analyzed (Participants) | 37 | 42 | 32
  Participants with Scale 6 at Day 4 | 0 | 1 | 0
  Participants with Scale 7 at Day 4: number analyzed (Participants) | 37 | 42 | 32
  Participants with Scale 7 at Day 4 | 1 | 0 | 0
  Participants with Scale 8 at Day 4: number analyzed (Participants) | 37 | 42 | 32
  Participants with Scale 8 at Day 4 | 0 | 0 | 0
  Participants with Scale 0 at Day 5: number analyzed (Participants) | 45 | 48 | 40
  Participants with Scale 0 at Day 5 | 0 | 1 | 0
  Participants with Scale 1 at Day 5: number analyzed (Participants) | 45 | 48 | 40
  Participants with Scale 1 at Day 5 | 9 | 6 | 6
  Participants with Scale 2 at Day 5: number analyzed (Participants) | 45 | 48 | 40
  Participants with Scale 2 at Day 5 | 4 | 5 | 4
  Participants with Scale 3 at Day 5: number analyzed (Participants) | 45 | 48 | 40
  Participants with Scale 3 at Day 5 | 13 | 18 | 16
  Participants with Scale 4 at Day 5: number analyzed (Participants) | 45 | 48 | 40
  Participants with Scale 4 at Day 5 | 11 | 14 | 14
  Participants with Scale 5 at Day 5: number analyzed (Participants) | 45 | 48 | 40
  Participants with Scale 5 at Day 5 | 6 | 3 | 0
  Participants with Scale 6 at Day 5: number analyzed (Participants) | 45 | 48 | 40
  Participants with Scale 6 at Day 5 | 0 | 1 | 0
  Participants with Scale 7 at Day 5: number analyzed (Participants) | 45 | 48 | 40
  Participants with Scale 7 at Day 5 | 2 | 0 | 0
  Participants with Scale 8 at Day 5: number analyzed (Participants) | 45 | 48 | 40
  Participants with Scale 8 at Day 5 | 0 | 0 | 0
  Participants with Scale 0 at Day 7: number analyzed (Participants) | 47 | 48 | 42
  Participants with Scale 0 at Day 7 | 0 | 1 | 1
  Participants with Scale 1 at Day 7: number analyzed (Participants) | 47 | 48 | 42
  Participants with Scale 1 at Day 7 | 15 | 16 | 15
  Participants with Scale 2 at Day 7: number analyzed (Participants) | 47 | 48 | 42
  Participants with Scale 2 at Day 7 | 11 | 9 | 8
  Participants with Scale 3 at Day 7: number analyzed (Participants) | 47 | 48 | 42
  Participants with Scale 3 at Day 7 | 10 | 14 | 11
  Participants with Scale 4 at Day 7: number analyzed (Participants) | 47 | 48 | 42
  Participants with Scale 4 at Day 7 | 4 | 5 | 7
  Participants with Scale 5 at Day 7: number analyzed (Participants) | 47 | 48 | 42
  Participants with Scale 5 at Day 7 | 5 | 2 | 0
  Participants with Scale 6 at Day 7: number analyzed (Participants) | 47 | 48 | 42
  Participants with Scale 6 at Day 7 | 0 | 1 | 0
  Participants with Scale 7 at Day 7: number analyzed (Participants) | 47 | 48 | 42
  Participants with Scale 7 at Day 7 | 2 | 0 | 0
  Participants with Scale 8 at Day 7: number analyzed (Participants) | 47 | 48 | 42
  Participants with Scale 8 at Day 7 | 0 | 0 | 0
  Participants with Scale 0 at Day 10: number analyzed (Participants) | 43 | 42 | 35
  Participants with Scale 0 at Day 10 | 5 | 2 | 2
  Participants with Scale 1 at Day 10: number analyzed (Participants) | 43 | 42 | 35
  Participants with Scale 1 at Day 10 | 16 | 21 | 18
  Participants with Scale 2 at Day 10: number analyzed (Participants) | 43 | 42 | 35
  Participants with Scale 2 at Day 10 | 8 | 4 | 7
  Participants with Scale 3 at Day 10: number analyzed (Participants) | 43 | 42 | 35
  Participants with Scale 3 at Day 10 | 5 | 10 | 7
  Participants with Scale 4 at Day 10: number analyzed (Participants) | 43 | 42 | 35
  Participants with Scale 4 at Day 10 | 5 | 2 | 1
  Participants with Scale 5 at Day 10: number analyzed (Participants) | 43 | 42 | 35
  Participants with Scale 5 at Day 10 | 2 | 2 | 0
  Participants with Scale 6 at Day 10: number analyzed (Participants) | 43 | 42 | 35
  Participants with Scale 6 at Day 10 | 0 | 1 | 0
  Participants with Scale 7 at Day 10: number analyzed (Participants) | 43 | 42 | 35
  Participants with Scale 7 at Day 10 | 1 | 0 | 0
  Participants with Scale 8 at Day 10: number analyzed (Participants) | 43 | 42 | 35
  Participants with Scale 8 at Day 10 | 1 | 0 | 0
  Participants with Scale 0 at Day 14: number analyzed (Participants) | 48 | 49 | 44
  Participants with Scale 0 at Day 14 | 5 | 5 | 6
  Participants with Scale 1 at Day 14: number analyzed (Participants) | 48 | 49 | 44
  Participants with Scale 1 at Day 14 | 26 | 25 | 23
  Participants with Scale 2 at Day 14: number analyzed (Participants) | 48 | 49 | 44
  Participants with Scale 2 at Day 14 | 7 | 8 | 8
  Participants with Scale 3 at Day 14: number analyzed (Participants) | 48 | 49 | 44
  Participants with Scale 3 at Day 14 | 5 | 6 | 7
  Participants with Scale 4 at Day 14: number analyzed (Participants) | 48 | 49 | 44
  Participants with Scale 4 at Day 14 | 2 | 3 | 0
  Participants with Scale 5 at Day 14: number analyzed (Participants) | 48 | 49 | 44
  Participants with Scale 5 at Day 14 | 0 | 1 | 0
  Participants with Scale 6 at Day 14: number analyzed (Participants) | 48 | 49 | 44
  Participants with Scale 6 at Day 14 | 1 | 1 | 0
  Participants with Scale 7 at Day 14: number analyzed (Participants) | 48 | 49 | 44
  Participants with Scale 7 at Day 14 | 0 | 0 | 0
  Participants with Scale 8 at Day 14: number analyzed (Participants) | 48 | 49 | 44
  Participants with Scale 8 at Day 14 | 2 | 0 | 0
  Participants with Scale 0 at Day 21: number analyzed (Participants) | 43 | 48 | 43
  Participants with Scale 0 at Day 21 | 8 | 8 | 7
  Participants with Scale 1 at Day 21: number analyzed (Participants) | 43 | 48 | 43
  Participants with Scale 1 at Day 21 | 22 | 30 | 35
  Participants with Scale 2 at Day 21: number analyzed (Participants) | 43 | 48 | 43
  Participants with Scale 2 at Day 21 | 9 | 7 | 1
  Participants with Scale 3 at Day 21: number analyzed (Participants) | 43 | 48 | 43
  Participants with Scale 3 at Day 21 | 1 | 0 | 0
  Participants with Scale 4 at Day 21: number analyzed (Participants) | 43 | 48 | 43
  Participants with Scale 4 at Day 21 | 0 | 2 | 0
  Participants with Scale 5 at Day 21: number analyzed (Participants) | 43 | 48 | 43
  Participants with Scale 5 at Day 21 | 0 | 0 | 0
  Participants with Scale 6 at Day 21: number analyzed (Participants) | 43 | 48 | 43
  Participants with Scale 6 at Day 21 | 0 | 1 | 0
  Participants with Scale 7 at Day 21: number analyzed (Participants) | 43 | 48 | 43
  Participants with Scale 7 at Day 21 | 1 | 0 | 0
  Participants with Scale 8 at Day 21: number analyzed (Participants) | 43 | 48 | 43
  Participants with Scale 8 at Day 21 | 2 | 0 | 0
  Participants with Scale 0 at Day 28: number analyzed (Participants) | 48 | 51 | 44
  Participants with Scale 0 at Day 28 | 14 | 11 | 15
  Participants with Scale 1 at Day 28: number analyzed (Participants) | 48 | 51 | 44
  Participants with Scale 1 at Day 28 | 24 | 35 | 24
  Participants with Scale 2 at Day 28: number analyzed (Participants) | 48 | 51 | 44
  Participants with Scale 2 at Day 28 | 5 | 3 | 4
  Participants with Scale 3 at Day 28: number analyzed (Participants) | 48 | 51 | 44
  Participants with Scale 3 at Day 28 | 2 | 1 | 0
  Participants with Scale 4 at Day 28: number analyzed (Participants) | 48 | 51 | 44
  Participants with Scale 4 at Day 28 | 1 | 0 | 1
  Participants with Scale 5 at Day 28: number analyzed (Participants) | 48 | 51 | 44
  Participants with Scale 5 at Day 28 | 0 | 0 | 0
  Participants with Scale 6 at Day 28: number analyzed (Participants) | 48 | 51 | 44
  Participants with Scale 6 at Day 28 | 0 | 0 | 0
  Participants with Scale 7 at Day 28: number analyzed (Participants) | 48 | 51 | 44
  Participants with Scale 7 at Day 28 | 0 | 0 | 0
  Participants with Scale 8 at Day 28: number analyzed (Participants) | 48 | 51 | 44
  Participants with Scale 8 at Day 28 | 2 | 1 | 0
  Participants with Scale 0 at Day 44: number analyzed (Participants) | 48 | 52 | 43
  Participants with Scale 0 at Day 44 | 17 | 17 | 22
  Participants with Scale 1 at Day 44: number analyzed (Participants) | 48 | 52 | 43
  Participants with Scale 1 at Day 44 | 23 | 30 | 20
  Participants with Scale 2 at Day 44: number analyzed (Participants) | 48 | 52 | 43
  Participants with Scale 2 at Day 44 | 4 | 4 | 1
  Participants with Scale 3 at Day 44: number analyzed (Participants) | 48 | 52 | 43
  Participants with Scale 3 at Day 44 | 2 | 0 | 0
  Participants with Scale 4 at Day 44: number analyzed (Participants) | 48 | 52 | 43
  Participants with Scale 4 at Day 44 | 0 | 0 | 0
  Participants with Scale 5 at Day 44: number analyzed (Participants) | 48 | 52 | 43
  Participants with Scale 5 at Day 44 | 0 | 0 | 0
  Participants with Scale 6 at Day 44: number analyzed (Participants) | 48 | 52 | 43
  Participants with Scale 6 at Day 44 | 0 | 0 | 0
  Participants with Scale 7 at Day 44: number analyzed (Participants) | 48 | 52 | 43
  Participants with Scale 7 at Day 44 | 0 | 0 | 0
  Participants with Scale 8 at Day 44: number analyzed (Participants) | 48 | 52 | 43
  Participants with Scale 8 at Day 44 | 2 | 1 | 0
  Participants with Scale 0 at Day 60: number analyzed (Participants) | 47 | 51 | 45
  Participants with Scale 0 at Day 60 | 18 | 17 | 22
  Participants with Scale 1 at Day 60: number analyzed (Participants) | 47 | 51 | 45
  Participants with Scale 1 at Day 60 | 24 | 31 | 22
  Participants with Scale 2 at Day 60: number analyzed (Participants) | 47 | 51 | 45
  Participants with Scale 2 at Day 60 | 3 | 2 | 1
  Participants with Scale 3 at Day 60: number analyzed (Participants) | 47 | 51 | 45
  Participants with Scale 3 at Day 60 | 0 | 0 | 0
  Participants with Scale 4 at Day 60: number analyzed (Participants) | 47 | 51 | 45
  Participants with Scale 4 at Day 60 | 0 | 0 | 0
  Participants with Scale 5 at Day 60: number analyzed (Participants) | 47 | 51 | 45
  Participants with Scale 5 at Day 60 | 0 | 0 | 0
  Participants with Scale 6 at Day 60: number analyzed (Participants) | 47 | 51 | 45
  Participants with Scale 6 at Day 60 | 0 | 0 | 0
  Participants with Scale 7 at Day 60: number analyzed (Participants) | 47 | 51 | 45
  Participants with Scale 7 at Day 60 | 0 | 0 | 0
  Participants with Scale 8 at Day 60: number analyzed (Participants) | 47 | 51 | 45
  Participants with Scale 8 at Day 60 | 2 | 1 | 0

7. Secondary Outcome: Time to Reach Peripheral Capillary Oxygen Saturation (SpO2) Greater Than or Equal to 94 Percent for at Least 24 Hours in Room Air
Description: SpO2 is an estimate of the amount of oxygen in the blood. It is the percentage of hemoglobin containing oxygen compared to the total amount of hemoglobin in the blood (that is, oxygenated hemoglobin versus oxygenated and non-oxygenated hemoglobin). SpO2 measured by pulse oximetry. The time to SPO2 greater than or equal to (>=) 94 percent (%) sustained for at least 24 hours in room air is reported in days.
Time Frame: Day 1 through Day 28
Population: Intent-to-Treat analysis set included all participants who had received at least one dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | M5049 50 Milligram (mg) | M5049 100 mg
Number analyzed (Participants) | 49 | 54 | 46
Days | 4.7 [2.8 to 6.9] | 4.8 [3.2 to 5.9] | 5.0 [3.9 to 9.0]

8. Secondary Outcome: Percentage of Participants With All-Cause Mortality
Description: Percentage of Participants who died for any reason reported.
Time Frame: Day 1 through Day 60
Population: Intent-to-Treat analysis set included all participants who had received at least one dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | M5049 50 Milligram (mg) | M5049 100 mg
Number analyzed (Participants) | 49 | 54 | 46
Percentage of participants | 4.1 [1.1 to 13.7] | 1.9 [0.3 to 9.8] | 0.0 [0.0 to 7.7]

9. Secondary Outcome: Time to Intensive Care Unit (ICU) Admission
Description: Time to ICU admission was defined as the time from first dose (Day 1) to the date/time of ICU admission, or death, whichever occurs first, in days. Event-free survival function for time to event (ICU admission or death) estimated via Kaplan-Meier method.
Time Frame: Day 1 through Day 28
Population: Intent-to-Treat analysis set included all participants who had received at least one dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | M5049 50 Milligram (mg) | M5049 100 mg
Number analyzed (Participants) | 49 | 54 | 46
Days | NA [NA to NA] — NA = Value not estimable (NE) due to an insufficient number of events | NA [NA to NA] — NA = Value not estimable (NE) due to an insufficient number of events | NA [NA to NA] — NA = Value not estimable (NE) due to an insufficient number of events

10. Secondary Outcome: Time to Non-Invasive Mechanical Ventilation
Description: Time to non-invasive mechanical ventilation was defined as the time from first dose (Day 1) to the date/time of clinical status >= 5, in days. Event-free survival function for time to event (Non-invasive mechanical ventilation or death) estimated via Kaplan-Meier method. Clinical status was based on data collected on the 'Ordinal Scale for Clinical Status and is assessed with the following ordinal scale: 0. Uninfected: no clinical or virological evidence of infection; 1. Ambulatory: no limitation of activities; 2. Ambulatory: limitation of activities; 3. Hospitalized, mild disease: hospitalized, no oxygen therapy; 4. Hospitalized, mild disease: oxygen by mask or nasal prongs; 5. Hospitalized, severe disease: noninvasive ventilation or high-flow oxygen; 6. Hospitalized, severe disease: intubation and mechanical ventilation; 7. Hospitalized, severe disease: ventilation plus additional organ support for example: vasopressors, and ECMO; 8. Death
Time Frame: Day 1 through Day 28
Population: Intent-to-Treat analysis set included all participants who had received at least one dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | M5049 50 Milligram (mg) | M5049 100 mg
Number analyzed (Participants) | 49 | 54 | 46
Days | NA [NA to NA] — NA = Value not estimable (NE) due to an insufficient number of events. | NA [NA to NA] — NA = Value not estimable (NE) due to an insufficient number of events. | NA [NA to NA] — NA = Value not estimable (NE) due to an insufficient number of events.

11. Secondary Outcome: Time to Invasive Mechanical Ventilation
Description: Time to invasive mechanical ventilation was defined as the time from first dose (Day 1) to the date/time of clinical status >= 6, in days. Event-free survival function for time to event (invasive mechanical ventilation or death) estimated via Kaplan-Meier method. Clinical status was based on data collected on the 'Ordinal Scale for Clinical Status and is assessed with the following ordinal scale: 0. Uninfected: no clinical or virological evidence of infection; 1. Ambulatory: no limitation of activities; 2. Ambulatory: limitation of activities; 3. Hospitalized, mild disease: hospitalized, no oxygen therapy; 4. Hospitalized, mild disease: oxygen by mask or nasal prongs; 5. Hospitalized, severe disease: noninvasive ventilation or high-flow oxygen; 6. Hospitalized, severe disease: intubation and mechanical ventilation; 7. Hospitalized, severe disease: ventilation plus additional organ support for example: vasopressors, and ECMO; 8. Death.
Time Frame: Day 1 through Day 28
Population: Intent-to-Treat analysis set included all participants who had received at least one dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | M5049 50 Milligram (mg) | M5049 100 mg
Number analyzed (Participants) | 49 | 54 | 46
Days | NA [NA to NA] — NA = Value not estimable (NE) due to an insufficient number of events. | NA [NA to NA] — NA = Value not estimable (NE) due to an insufficient number of events. | NA [NA to NA] — NA = Value not estimable (NE) due to an insufficient number of events.

12. Secondary Outcome: Total Length of Stay in Intensive Care Unit (ICU)
Description: Total days in the ICU was defined as the sum, for all ICU admissions, of the time from ICU admission to the date of ICU discharge, in days.
Time Frame: Day 1 through Day 60
Population: Intent-to-Treat analysis set included all participants who had received at least one dose of study intervention.
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo | M5049 50 Milligram (mg) | M5049 100 mg
Number analyzed (Participants) | 49 | 54 | 46
Days | 7.1 [1 to 17] | 10.2 [3 to 23] | 3.7 [2 to 6]

13. Secondary Outcome: Total Length of Hospitalization Stay
Description: Total days in the hospital was defined as the sum, for all hospitalization events, of the time from first dose to the date of hospital discharge in days.
Time Frame: Day 1 through Day 60
Population: Intent-to-Treat analysis set included all participants who had received at least one dose of study intervention.
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo | M5049 50 Milligram (mg) | M5049 100 mg
Number analyzed (Participants) | 49 | 54 | 46
Days | 7.0 [2 to 41] | 6.0 [2 to 29] | 6.0 [2 to 17]

14. Secondary Outcome: Time to Hospital Discharge
Description: The time to hospital discharge, defined as the time from first dose (Day 1) to the date of first hospitalization discharge, in days.
Time Frame: Day 1 through Day 60
Population: Intent-to-Treat analysis set included all participants who had received at least one dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | M5049 50 Milligram (mg) | M5049 100 mg
Number analyzed (Participants) | 49 | 54 | 46
Days | 5.1 [3.7 to 6.0] | 5.1 [4.0 to 7.1] | 4.7 [3.7 to 5.9]

15. Secondary Outcome: Percent Change From Baseline in Inflammatory Biomarkers Over Time
Description: C-Reactive Protein, D-Dimer and Ferritin inflammatory biomarkers were analyzed for this study. Percent Change From Baseline in Inflammatory Biomarkers Over Time were reported here.
Time Frame: Baseline, Day 3, Day7, Day 10, Day 14 and Day 28
Population: Pharmacodynamics (PD) analysis set included all participants who received atleast 1 dose of study intervention, for whom atleast 1 postbaseline serum biomarker was obtained without any relevant protocol deviations or events that may have an influence on PD. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and Number Analyzed" signified those participants who were evaluable for the specified category at given time points.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | M5049 50 Milligram (mg) | M5049 100 mg
Number analyzed (Participants) | 41 | 39 | 35
Percent change
  Percent change at Day 3 in C-Reactive Protein: number analyzed (Participants) | 41 | 37 | 35
  Percent change at Day 3 in C-Reactive Protein | -0.8 (113.57) | 48.2 (399.18) | -45.1 (59.64)
  Percent change at Day 7 in C-Reactive Protein: number analyzed (Participants) | 30 | 38 | 29
  Percent change at Day 7 in C-Reactive Protein | -48.1 (69.03) | -50.4 (133.43) | -74.3 (32.19)
  Percent change at Day 10 in C-Reactive Protein: number analyzed (Participants) | 19 | 17 | 14
  Percent change at Day 10 in C-Reactive Protein | 10.5 (182.35) | -58.2 (43.93) | -68.3 (81.09)
  Percent change at Day 14 in C-Reactive Protein: number analyzed (Participants) | 37 | 39 | 33
  Percent change at Day 14 in C-Reactive Protein | -62.1 (39.95) | 24.6 (543.06) | -51.2 (159.45)
  Percent change at Day 28 in C-Reactive Protein: number analyzed (Participants) | 28 | 33 | 31
  Percent change at Day 28 in C-Reactive Protein | -62.0 (91.47) | -27.0 (253.69) | -72.4 (45.01)
  Percent change at Day 3 in D-Dimer: number analyzed (Participants) | 37 | 35 | 29
  Percent change at Day 3 in D-Dimer | 62.5 (150.19) | 2008.7 (11813.54) | 2093.9 (11278.04)
  Percent change at Day 7 in D-Dimer: number analyzed (Participants) | 29 | 35 | 26
  Percent change at Day 7 in D-Dimer | 184.5 (517.94) | 35.4 (197.99) | 1922.7 (9449.18)
  Percent change at Day 10 in D-Dimer: number analyzed (Participants) | 17 | 12 | 10
  Percent change at Day 10 in D-Dimer | 2004.2 (5139.01) | 62.6 (202.41) | 171.3 (501.83)
  Percent change at Day 14 in D-Dimer: number analyzed (Participants) | 36 | 39 | 30
  Percent change at Day 14 in D-Dimer | 1136.7 (6760.10) | 0.7 (86.62) | 15.1 (100.97)
  Percent change at Day 28 in D-Dimer: number analyzed (Participants) | 27 | 30 | 25
  Percent change at Day 28 in D-Dimer | 893.4 (4731.82) | -5.9 (61.09) | 1371.6 (6985.20)
  Percent change at Day 3 in Ferritin: number analyzed (Participants) | 35 | 35 | 29
  Percent change at Day 3 in Ferritin | 17.8 (83.23) | 3.4 (43.05) | -7.2 (20.63)
  Percent change at Day 7 in Ferritin: number analyzed (Participants) | 29 | 38 | 25
  Percent change at Day 7 in Ferritin | 11.1 (151.34) | -22.7 (40.53) | -19.8 (27.64)
  Percent change at Day 10 in Ferritin: number analyzed (Participants) | 15 | 17 | 11
  Percent change at Day 10 in Ferritin | 21.4 (167.00) | -25.4 (31.52) | -39.7 (25.13)
  Percent change at Day 14 in Ferritin: number analyzed (Participants) | 33 | 37 | 30
  Percent change at Day 14 in Ferritin | -29.4 (117.71) | -47.8 (31.56) | -49.9 (18.54)
  Percent change at Day 28 in Ferritin: number analyzed (Participants) | 25 | 32 | 27
  Percent change at Day 28 in Ferritin | -61.3 (35.83) | -62.3 (25.83) | -63.2 (15.71)

16. Secondary Outcome: Percent Change From Baseline in Serum Cytokine Biomarkers
Description: Interleukin 6 and Interleukin 8 serum cytokine biomarkers were analyzed. Percent Change From Baseline in Serum Cytokine Biomarkers were reported.
Time Frame: Baseline, Day 3, Day7, Day 14 and Day 28
Population: PD analysis set included all participants who received at least 1 dose of study intervention, for whom at least 1 postbaseline serum biomarker was obtained without any relevant protocol deviations or events that may have an influence on PD. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and Number Analyzed" signified those participants who were evaluable for the specified category at given time points.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | M5049 50 Milligram (mg) | M5049 100 mg
Number analyzed (Participants) | 38 | 38 | 35
Percent change
  Percent change at Day 3 in Interleukin 6: number analyzed (Participants) | 38 | 34 | 35
  Percent change at Day 3 in Interleukin 6 | 51.2 (257.64) | -17.8 (38.95) | 1722.3 (10240.47)
  Percent change at Day 7 in Interleukin 6: number analyzed (Participants) | 30 | 33 | 29
  Percent change at Day 7 in Interleukin 6 | 35.2 (167.99) | 1.1 (159.45) | -25.5 (42.41)
  Percent change at Day 14 in Interleukin 6: number analyzed (Participants) | 37 | 38 | 35
  Percent change at Day 14 in Interleukin 6 | 20.2 (164.19) | 55.2 (476.42) | 275.1 (1745.50)
  Percent change at Day 28 in Interleukin 6: number analyzed (Participants) | 32 | 32 | 33
  Percent change at Day 28 in Interleukin 6 | -21.0 (41.33) | -27.3 (37.78) | -30.1 (36.93)
  Percent change at Day 3 in Interleukin 8: number analyzed (Participants) | 38 | 34 | 35
  Percent change at Day 3 in Interleukin 8 | 42.5 (165.56) | 2.0 (77.66) | 126.6 (574.74)
  Percent change at Day 7 in Interleukin 8: number analyzed (Participants) | 30 | 33 | 29
  Percent change at Day 7 in Interleukin 8 | 923.4 (4432.63) | 60.2 (253.12) | 28.5 (113.48)
  Percent change at Day 14 in Interleukin 8: number analyzed (Participants) | 37 | 38 | 35
  Percent change at Day 14 in Interleukin 8 | 408.9 (1776.87) | 35.4 (147.85) | 283.5 (1616.08)
  Percent change at Day 28 in Interleukin 8: number analyzed (Participants) | 32 | 32 | 33
  Percent change at Day 28 in Interleukin 8 | -4.3 (90.29) | -13.0 (59.00) | -1.8 (123.62)

17. Secondary Outcome: Percentage of Participants With Relapse
Description: Relapse refers to rehospitalization due to worsening oxygenation, with either a positive result of any respiratory pathogenic nucleic acid test, or worsening lesions on chest imaging.
Time Frame: Day 5 through Day 60
Population: Intent-to-Treat analysis set included all participants who had received at least one dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | M5049 50 Milligram (mg) | M5049 100 mg
Number analyzed (Participants) | 49 | 54 | 46
Percentage of participants | 0.0 [0.00 to 7.27] | 0.0 [0.00 to 6.64] | 0.0 [0.00 to 7.71]

18. Secondary Outcome: Percentage of Participants Who Are Re-Hospitalized
Description: Percentage or participants who are re-hospitalized due to coronavirus disease 2019 (Covid-19) complications were reported.
Time Frame: Day 5 through Day 60
Population: Intent-to-Treat analysis set included all participants who had received at least one dose of study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | M5049 50 Milligram (mg) | M5049 100 mg
Number analyzed (Participants) | 49 | 54 | 46
Percentage of participants | 0.0 [0.00 to 7.27] | 0.0 [0.00 to 6.76] | 2.2 [0.38 to 11.34]

ADVERSE EVENTS:
Time Frame: Baseline up to Day 60
Arm/Group | Placebo | M5049 50 Milligram (mg) | M5049 100 mg
All-Cause Mortality (participants affected / at risk) | 2/49 | 1/54 | 0/46
Serious Adverse Events (participants affected / at risk) | 9/49 | 5/54 | 1/46
Other Adverse Events (participants affected / at risk) | 12/49 | 15/54 | 10/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=49) | M5049 50 Milligram (mg) (N=54) | M5049 100 mg (N=46)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 3 | 4 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0
Oxygen saturation decreased (Investigations) | 2 | 0 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=49) | M5049 50 Milligram (mg) (N=54) | M5049 100 mg (N=46)
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 3
Constipation (Gastrointestinal disorders) | 2 | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 0
Alanine aminotransferase increased (Investigations) | 6 | 1 | 1
Transaminases increased (Investigations) | 1 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3 | 4
Insomnia (Psychiatric disorders) | 4 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT04448756/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/56/NCT04448756/SAP_001.pdf